CLINICAL TRIAL: NCT01090908
Title: A Multi-Center, Open Label Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Ciprofloxacin For Inhalation (CFI) Given Daily For 14 Days To Stable Cystic Fibrosis Patients Ages 6 To 17 With Pseudomonas Aeruginosa
Brief Title: Evaluation of Ciprofloxacin for Inhalation to Cystic Fibrosis Patients With P. Aeruginosa
Status: Withdrawn | Type: Observational
Sponsor: Aradigm Corporation (Industry)
Responsible Party: David E. Geller, M.D., Nemours Children's Clinic
Organization: Savara Inc. (Industry)
Other Study IDs: ARD-3100-1001
Record Dates: First submitted 2010-03-11; First posted 2010-03-23 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2012-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ages 6-11 years
  Interventions: Drug: Antibiotic
- Ages 12-17 years
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic

SUMMARY:
This is a Phase 1/2a, multicenter study, designed to evaluate the pharmacokinetics, safety, and tolerability of once daily administration of 150 mg of Ciprofloxacin for Inhalation (CFI) in patients with Cystic Fibrosis who have a history of chronic P. aeruginosa lung infection.

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter study, designed to evaluate the pharmacokinetics, safety, and tolerability of once daily administration of 150 mg of Ciprofloxacin for Inhalation (CFI) in patients with Cystic Fibrosis who have a history of chronic P. aeruginosa lung infection. Patients will be enrolled and followed in this study for 1 month. This study will consist of a Screening Phase, a Treatment Phase consisting of a 14 days, and a Follow up Phase consisting of a 14 days Off-treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 17 years of age (inclusive) at Visit 1.
* Positive sputum culture for P. aeruginosa
* Clinical diagnosis of CF
* FEV1 greater than or equal to 40% predicted normal lung function
* Able to perform spirometry testing reproducibly according to ATS guidelines.

Exclusion Criteria:

* Use of an investigational agent within 30 days prior to Visit 1 (first dosing visit).
* History of sputum culture or deep-throat cough swab (or BAL) culture yielding Burkholderia cepacia (B. cepacia), within 2 years prior to screening and/or sputum culture yielding B. cepacia at the Screening visit;
* Use of any nebulized or systemic antibiotics within 14 days prior to Visit 1, other than maintenance oral macrolides that has been consistently used for at least 28 days prior to Visit 1.
* History of intolerance or hypersensitivity to quinolone or fluoroquinolone class antibiotics
* History of lung transplantation.
* AST, ALT or total bilirubin > 3 x upper limit of normal at screening.
* History of hemoptysis > 30 cc per episode during the 28 days prior to Visit 1.
* Other present conditions, abnormality in screening laboratory tests or physical examination findings, that in the opinion of the Investigator or Medical Monitor would compromise the safety of the patient or the quality of the data.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatrics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Serum pharmacokinetics | Day 1

SECONDARY OUTCOMES:
Microbiological efficacy | Day 14
Changes in spirometry | Days 1, 7, 14
Quality of life (CFQ-R) | Days 1, 7, 14

CONTACTS AND LOCATIONS:
Overall Officials: P Bruinenber, MD, Study Director — Aradigm Corporation